CLINICAL TRIAL: NCT00961155
Title: Usefulness of Exhaled Breath Condensate and FENO for Evaluation of Markers of Airway Inflammation in Children With Asthma
Brief Title: Usefulness of Exhaled Breath Condensate for Evaluation of Markers of Airway Inflammation in Children With Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Professor, Medical University of Lodz
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RNN/137/08/KE
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: asthma; children; EBC; exposure to tabacco; antiasthma treatment
MeSH Terms: conditions — Asthma | interventions — ciclesonide; montelukast; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- cyklezonid (Active Comparator): children will receive 160 mcg once daily cyklezonid for 3 months
  Interventions: Drug: cyklezonid
- montelukast sodium (Active Comparator): children will receive 5 or 10 mg montelukast sodium for 3 months
  Interventions: Drug: montelukast sodium
- placebo (Placebo Comparator): children will receive placebo for 8 weeks out of allergy season to house dust mite
  Interventions: Drug: placebo
- formoterol (Active Comparator): children will receive formoterol aerolzol 12mcg twice daily for 3 months
  Interventions: Drug: formoterol 12 mcg twice daily

INTERVENTIONS:
Drug: cyklezonid — 160 mcg once daily
  Other Names: Alvesco
  Arms: cyklezonid
Drug: montelukast sodium — 5 or 10 mg according to age once daily
  Arms: montelukast sodium
Drug: placebo — fluticasone placebo twice daily, montelukast placebo once daily
  Arms: placebo
Drug: formoterol 12 mcg twice daily — formoterol 12 mcg twice daily will be given to children for 3 months
  Other Names: Formoterol
  Arms: formoterol

SUMMARY:
Exhaled breath condensate (EBC) has emerged as a novel noninvasive technique for assessment of airway inflammation, and it provides information on airway lining fluid composition. Traditionally, such assessment relies on invasive diagnostic tools such as bronchial biopsy and bronchoalveolar lavage (BAL) to obtain specimens from the airway but it is very uncomfortable procedure especially for young patients. The aim of this study is to evaluate the effect of allergic disease, disease monitoring and exposure to tobacco smoke on airway inflammation measured by markers in exhaled breath condensate (EBC) in children with asthma allergic to house dust mite. Also, we aim to assess correlations between cytokine concentrations in EBC and clinical characteristic of the patients with exercise-induced bronchoconstriction as another phenotype of asthma.

DETAILED DESCRIPTION:
Markers that can be identified in the EBC of patients with asthma include pH, hydrogen peroxide, nitrogen oxides, eicosanoids, isoprostanes, adenosine, certain cytokines, chemokines, and growth factors. Concentrations of these biomarkers are influenced by inflammation, oxidative stress, and can be modulated by therapeutic interventions. There is evidence that some markers in EBC differ between patients with asthma and controls, and some of them can correlate with asthma severity score, lung function. The aim of this study is to evaluate the effect of allergic disease, disease monitoring and exposure to tobacco smoke on airway inflammation measured by markers in exhaled breath condensate (EBC) in children with asthma allergic to house dust mite. We will also evaluate the effect of antiasthmatic treatment applied out of dust season on the number of exacerbations in "asthma epidemic" in September. We will evaluate the effect of exposure to tobacco smoke on antiasthmatic treatment.

Also, we aim to assess correlations between cytokine concentrations in EBC and clinical characteristic of the patients with exercise-induced bronchoconstriction (EIB) as another phenotype of asthma. At the first study vist patients with EIB underwent fractional exhaled nitric oxide measurement (FeNO) and baseline spirometry, performed exercise treadmill challenge (ETC) and EBC samples were obtained at the end of ETC.

ELIGIBILITY:
Inclusion Criteria:

* children with mild to moderate asthma allergic to house dust mite exposed/nonexposed to tobacco smoke
* healthy children

Exclusion Criteria:

* sensitization to allergens other than house dust mites
* other chronic diseases
* asthma exacerbation
* pregnancy
* oral corticosteroids for 4 weeks before the study
* montelukast sodium for 2 weeks before the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of IL-4, 5, 6, 8, 16, MIG, TNF- alpha, MCP-1 in EBC. Measurement of ECP, eosinophil blood count, cotinine and total IgE in blood. | visit 1-6

SECONDARY OUTCOMES:
Measurement of FENO, bronchial hyperreactivity, exercise treadmill challenge, lung function and clinical evaluation | visits 1-6

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Jerzynska, MD PhD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD PhD Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Agnieszka Brzozowska, MD, PhD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Poland, Lodz, Łódź Voivodeship, Poland